CLINICAL TRIAL: NCT01282658
Title: Genetic Variants and the Efficacy or Severe Adverse Reactions of CPT-11 Based Regimens in mCRC
Brief Title: Pharmacogenomics Study of CPT-11 as the First-line Chemotherapy for mCRC
Acronym: PSIFL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Wuhan University (Other)
Responsible Party: Yuan Xianglin, Tongji Hospital of Tongji Medical College, Hua Zhong University of Science & Technology
Other Study IDs: TJCC-001
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2010-11

CONDITIONS: Colorectal Cancer
Keywords: CPT-11,pharmacogenomics,colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colorectal cancer

SUMMARY:
Irinotecan (CPT-11) is now widely used as the first-line chemotherapy for mCRC. There were 4 key enzymes for CPT-11 metabolizing, CYP3A4, UDP-glucuronosyltransferase, carboxylesterase(CES), and ATP-binding cassette (ABC) transporters. Genetic variations of those enzymes may cause the heterogeneity in safety and efficacy of CPT-11. The aim of this study is to figure out the correlation between the genetic polymorphism and the drug response.

DETAILED DESCRIPTION:
collect blood samples,determining genetic contribution to the safety and efficacy of CPT-11.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal cancer
2. ≥ 18 years old
3. Measurable disease, defined as to RECIST criteria
4. Unresectable metastatic disease OR First recurrence/metastasis after adjuvant therapy and not suitable for operation
5. FOLFIRI±cetuximab/bevacizumab as the first-line therapy
6. Without expected course of radiotherapy during the first-line chemotherapy
7. No previous CPT-11 chemotherapy
8. ECOG performance status (PS) 0-2
9. Not pregnant or nursing and Negative pregnancy test
10. Voluntarily signed the informed consent
11. Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
12. AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN if f liver metastases present)
13. Creatinine clearance > 50 mL/min OR serum creatinine ≤ 1.5 times ULN

Exclusion Criteria:

1. Brain metastases with obvious symptoms
2. Severe bone marrow failure and can not be corrected
3. Chronic diarrhea history
4. Bowel obstruction without control
5. Mental illness without control
6. Clinically significant (i.e., active) cardiovascular disease, including any of the following: Cerebrovascular accidents/ Myocardial infarction/ Unstable angina/ New York Heart Association class II-IV congestive heart failure/ Serious cardiac arrhythmia requiring medication/ Uncontrolled hypertension
7. Other co-existing malignancy or malignancy diagnosed within the past 5 years, except for basal cell or squamous cell carcinoma, or carcinoma in situ of the cervix
8. Pelvic radiotherapy for the past 1 year
9. Known allergy to any of the components of the study medications
10. Serious, nonhealing wound or ulcer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-12 (Estimated); Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yuan X Lin, PHD, Principal Investigator — Tongji Hospital of Tongji Medical College, Hua Zhong University of Science & Technology
Locations (1):
- Tongji Hospital of Tongji Medical College, Hua Zhong University of Science & Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Van Cutsem E, Nordlinger B, Adam R, Kohne CH, Pozzo C, Poston G, Ychou M, Rougier P; European Colorectal Metastases Treatment Group. Towards a pan-European consensus on the treatment of patients with colorectal liver metastases. Eur J Cancer. 2006 Sep;42(14):2212-21. doi: 10.1016/j.ejca.2006.04.012. Epub 2006 Aug 10. PMID 16904315
- [Background] A Report of Cancer Incidence and Mortality from 34 Cancer Registries in China，2006. China Cancer 19:356-65, 2010
- [Background] Yoo PS, Lopez-Soler RI, Longo WE, Cha CH. Liver resection for metastatic colorectal cancer in the age of neoadjuvant chemotherapy and bevacizumab. Clin Colorectal Cancer. 2006 Sep;6(3):202-7. doi: 10.3816/CCC.2006.n.036. PMID 17026789
- [Background] Saltz LB, Cox JV, Blanke C, Rosen LS, Fehrenbacher L, Moore MJ, Maroun JA, Ackland SP, Locker PK, Pirotta N, Elfring GL, Miller LL. Irinotecan plus fluorouracil and leucovorin for metastatic colorectal cancer. Irinotecan Study Group. N Engl J Med. 2000 Sep 28;343(13):905-14. doi: 10.1056/NEJM200009283431302. PMID 11006366
- [Background] Douillard JY, Cunningham D, Roth AD, Navarro M, James RD, Karasek P, Jandik P, Iveson T, Carmichael J, Alakl M, Gruia G, Awad L, Rougier P. Irinotecan combined with fluorouracil compared with fluorouracil alone as first-line treatment for metastatic colorectal cancer: a multicentre randomised trial. Lancet. 2000 Mar 25;355(9209):1041-7. doi: 10.1016/s0140-6736(00)02034-1. PMID 10744089
- [Background] Rhodes KE, Zhang W, Yang D, Press OA, Gordon M, Vallbohmer D, Schultheis AM, Lurje G, Ladner RD, Fazzone W, Iqbal S, Lenz HJ. ABCB1, SLCO1B1 and UGT1A1 gene polymorphisms are associated with toxicity in metastatic colorectal cancer patients treated with first-line irinotecan. Drug Metab Lett. 2007 Jan;1(1):23-30. doi: 10.2174/187231207779814328. PMID 19356014
- [Background] Innocenti F, Undevia SD, Iyer L, Chen PX, Das S, Kocherginsky M, Karrison T, Janisch L, Ramirez J, Rudin CM, Vokes EE, Ratain MJ. Genetic variants in the UDP-glucuronosyltransferase 1A1 gene predict the risk of severe neutropenia of irinotecan. J Clin Oncol. 2004 Apr 15;22(8):1382-8. doi: 10.1200/JCO.2004.07.173. Epub 2004 Mar 8. PMID 15007088
- [Background] Ramchandani RP, Wang Y, Booth BP, Ibrahim A, Johnson JR, Rahman A, Mehta M, Innocenti F, Ratain MJ, Gobburu JV. The role of SN-38 exposure, UGT1A1*28 polymorphism, and baseline bilirubin level in predicting severe irinotecan toxicity. J Clin Pharmacol. 2007 Jan;47(1):78-86. doi: 10.1177/0091270006295060. PMID 17192505
- [Background] Marcuello E, Altes A, Menoyo A, Del Rio E, Gomez-Pardo M, Baiget M. UGT1A1 gene variations and irinotecan treatment in patients with metastatic colorectal cancer. Br J Cancer. 2004 Aug 16;91(4):678-82. doi: 10.1038/sj.bjc.6602042. PMID 15280927
- [Background] Carlini LE, Meropol NJ, Bever J, Andria ML, Hill T, Gold P, Rogatko A, Wang H, Blanchard RL. UGT1A7 and UGT1A9 polymorphisms predict response and toxicity in colorectal cancer patients treated with capecitabine/irinotecan. Clin Cancer Res. 2005 Feb 1;11(3):1226-36. PMID 15709193
- [Background] Mathijssen RH, Marsh S, Karlsson MO, Xie R, Baker SD, Verweij J, Sparreboom A, McLeod HL. Irinotecan pathway genotype analysis to predict pharmacokinetics. Clin Cancer Res. 2003 Aug 15;9(9):3246-53. PMID 12960109
- [Background] Ando Y, Hasegawa Y. Clinical pharmacogenetics of irinotecan (CPT-11). Drug Metab Rev. 2005;37(3):565-74. doi: 10.1080/03602530500316254. PMID 16257834
- [Background] Paradiso A, Xu J, Mangia A, Chiriatti A, Simone G, Zito A, Montemurro S, Giuliani F, Maiello E, Colucci G. Topoisomerase-I, thymidylate synthase primary tumour expression and clinical efficacy of 5-FU/CPT-11 chemotherapy in advanced colorectal cancer patients. Int J Cancer. 2004 Aug 20;111(2):252-8. doi: 10.1002/ijc.20208. PMID 15197779
- [Background] Braun MS, Richman SD, Quirke P, Daly C, Adlard JW, Elliott F, Barrett JH, Selby P, Meade AM, Stephens RJ, Parmar MK, Seymour MT. Predictive biomarkers of chemotherapy efficacy in colorectal cancer: results from the UK MRC FOCUS trial. J Clin Oncol. 2008 Jun 1;26(16):2690-8. doi: 10.1200/JCO.2007.15.5580. PMID 18509181
- [Background] Smith NF, Figg WD, Sparreboom A. Pharmacogenetics of irinotecan metabolism and transport: an update. Toxicol In Vitro. 2006 Mar;20(2):163-75. doi: 10.1016/j.tiv.2005.06.045. Epub 2005 Nov 3. PMID 16271446
- [Background] Hoskins JM, Marcuello E, Altes A, Marsh S, Maxwell T, Van Booven DJ, Pare L, Culverhouse R, McLeod HL, Baiget M. Irinotecan pharmacogenetics: influence of pharmacodynamic genes. Clin Cancer Res. 2008 Mar 15;14(6):1788-96. doi: 10.1158/1078-0432.CCR-07-1472. PMID 18347181
- [Derived] Yu Q, Zhang T, Xie C, Qiu H, Liu B, Huang L, Peng P, Feng J, Chen J, Zang A, Yuan X. UGT1A polymorphisms associated with worse outcome in colorectal cancer patients treated with irinotecan-based chemotherapy. Cancer Chemother Pharmacol. 2018 Jul;82(1):87-98. doi: 10.1007/s00280-018-3595-7. Epub 2018 May 4. PMID 29728798
- [Derived] Li J, Yu Q, Fu S, Xu M, Zhang T, Xie C, Feng J, Chen J, Zang A, Cai Y, Fu Q, Liu S, Zhang M, Hong Q, Huang L, Yuan X. A novel genetic score model of UGT1A1 and TGFB pathway as predictor of severe irinotecan-related diarrhea in metastatic colorectal cancer patients. J Cancer Res Clin Oncol. 2016 Jul;142(7):1621-8. doi: 10.1007/s00432-016-2176-6. Epub 2016 May 9. PMID 27160286
- [Derived] Huang L, Zhang T, Xie C, Liao X, Yu Q, Feng J, Ma H, Dai J, Li M, Chen J, Zang A, Wang Q, Ge S, Qin K, Cai J, Yuan X. SLCO1B1 and SLC19A1 gene variants and irinotecan-induced rapid response and survival: a prospective multicenter pharmacogenetics study of metastatic colorectal cancer. PLoS One. 2013 Oct 15;8(10):e77223. doi: 10.1371/journal.pone.0077223. eCollection 2013. PMID 24143213